CLINICAL TRIAL: NCT03541122
Title: Three Novel Radiological Indicators for Diagnosis of Adult Acetabular Dysplasia: a Self-controlled, Diagnostic Trial
Brief Title: Three Novel Radiological Indicators for Diagnosis of Adult Acetabular Dysplasia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Principal Investigator, Di Qin, Principal Investigator, Hebei Medical University Third Hospital
Other Study IDs: HebeiMUth-003
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Acetabular Dysplasia
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Patients will undergo pelvic X-ray examinations. Measurement indicators will include OFI, MUI, TBOI, CE angle, Sharp angle and AHI of the affected and healthy femoral heads. The investigators will determine the sensitivity and specificity of OFI, MUI and TBOI for the diagnosis of adult acetabular dysplasia, and compare the accuracy of diagnosis between these three indicators and CE angle, sharp angle, and AHI. Further analysis of risk factors for hip function will be implemented.
  Interventions: Diagnostic Test: pelvic X-ray examinations

INTERVENTIONS:
Diagnostic Test: pelvic X-ray examinations — Measurement indicators will include OFI, MUI, TBOI, CE angle, Sharp angle and AHI of the affected and healthy femoral heads.

SUMMARY:
Acetabular dysplasia often accompanies by acetabular bone hyperplasia and osteonecrosis of the femoral head. These pathological changes can alter the position of the center of the femoral head. Thus, measurement errors will be generated on the anteroposterior radiographs of the adult pelvis involving centre-edge angle, acetabular angle (Sharp angle), and acetabular head index, eventually resulting in the inaccurate diagnosis of acetabular dysplasia. Herein, the investigators describe the protocol to verify three novel X-ray indicators, including offshoring index (OFI), moving up index (MUI) and teardrop baseline offshoring index (TBOI) of the femoral head. All data will be expressed as relative ratios, as the investigators expect to make an accurate diagnosis through avoiding the generation of errors resulting from measurement angles.

DETAILED DESCRIPTION:
Acetabular dysplasia is a developmental malformation of the hip joint where the acetabulum become shallow and cannot fully cover the femoral head and the centre of the hip joint moves outward, resulting in an increased risk for joint subluxation or dislocation.

Current diagnosis of acetabular dysplasia mainly depends on the pelvic anteroposterior X-ray film to understand whether there is dislocation of the hip joint, whether the concentricity of the femoral head and acetabulum is consistent, and whether there is secondary osteoarthritis or other hip diseases, such as femoral head ischemic necrosis, hip joint tuberculosis, and rheumatoid arthritis. The commonly used measurement indicators include centre-edge (CE) angle, acetabular angle (Sharp angle), and acetabular head index (AHI). Moreover, some differences exist in the measurement results between male and female patients. Acetabular dysplasia often accompanies by acetabular bone hyperplasia and necrosis of the femoral head, which have a greater impact on radiographic measurements, especially when measured with angles. It is difficult to determine the radiological landmark for the lateral edge of the acetabular roof due to the existence of bone hyperplasia, which produces a great influence on the accuracy of the measurement of the centre-edge angle and Sharp angle.

ELIGIBILITY:
Inclusion Criteria:

* No experience in hip replacement, pelvic fixation or external fixation, and proximal femoral surgery;
* No marked pelvic tilt;
* No hip dislocation;
* No obvious hip deformity, such as significant collapse of the femoral head and severe hip traumatic arthritis;
* No significant lesions in the pelvis or proximal femur;
* Aged over 16 years;
* Provision of written informed consent.

Exclusion Criteria:

* Those with advanced osteoarthritis;
* Those with osteoarthritis secondary to acetabular dysplasia;
* Those with ankylosing spondylitis involving the hip joint;
* Those with rheumatoid arthritis;
* Those with inflammatory inflammation of the hip joint;
* Those with tumor lesions in the hip joint.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Potential patients will be informed of the study details through an announcement issued through the bulletin board of the Third Hospital of Hebei Medical University. Interested patients will directly contact the principle investigator via telephone, and among them, eligible patients will be required to provide written consent prior to the participation in the trial.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of offshoring index (OFI) | One day after hospitalization
  The sensitivity represents the percentage of actual patients who are correctly diagnosed with a disease. A higher sensitivity indicates a higher rate of correct diagnosis for acetabular dysplasia.

SECONDARY OUTCOMES:
The specificity of OFI,MUI and TBOI | One day after hospitalization
  The specificity represents the percentage of disease-free patients who are correctly diagnosed with no disease. A higher specificity indicates a higher rate of correct diagnosis for acetabular dysplasia.
The positive predictive value of OFI,MUI and TBOI | One day after hospitalization
  The positive predictive value represents the probability that the patient actually suffer from the disease (true positive rate) in all positive cases.
The negative predictive value of OFI,MUI and TBOI | One day after hospitalization
  The negative predictive value represents the probability that the patient does not suffer from have the disease. This value is often influenced by the sensitivity, specificity, and prevalence in all cases.
The positive likelihood ratio of OFI,MUI and TBOI | One day after hospitalization
  The positive likelihood ratio represents the probability of a patient who has the disease testing positive divided by the probability of a patient who does not have the disease testing positive.
The negative likelihood ratio of OFI,MUI and TBOI | One day after hospitalization
  The negative likelihood ratio represents the probability of a patient who has the disease testing negative divided by the probability of a patient who does not have the disease testing negative.

CONTACTS AND LOCATIONS:
Overall Officials: Di Qin, M.S., Principal Investigator — Third Hospital of Hebei Medical University
Locations (1):
- Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided